CLINICAL TRIAL: NCT02064231
Title: A Clinical Investigation Examining the Performance and Handling of New 2-piece Ostomy Products in 28 People With an Ileostomy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CP222
Record Dates: First submitted 2014-02-13; First posted 2014-02-17 (Estimated); Results first posted 2014-04-04 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-08

CONDITIONS: Ileostomy - Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coloplast Test A, Coloplast Test B, Own product (Experimental): The subjects first test Coloplast Test A and thereafter Coloplast Test B and finally their own product for 14 days
  Interventions: Device: Coloplast Test A; Device: Coloplast Test B; Device: Own product
- Coloplast Test C , Coloplast Test D, Own product (Experimental): The subjects first test Coloplast Test C and thereafter Coloplast Test D and finally their own product for 14 days
  Interventions: Device: Own product; Device: Coloplast Test C; Device: Coloplast Test D

INTERVENTIONS:
Device: Coloplast Test A — Coloplast Test A is a new ostomy appliance developed by Coloplast A/S
  Arms: Coloplast Test A, Coloplast Test B, Own product
Device: Coloplast Test B — Coloplast Test B is a newly developed ostomy appliance developed by Coloplast A/S
  Arms: Coloplast Test A, Coloplast Test B, Own product
Device: Own product — Own product is tested to get baseline results. Own product can be any 2-piece product that is commercially available. The manufactures can be Coloplast, Hollister, Convatec, Dansac, B. Braun and others.
Device: Coloplast Test C — Coloplast Test C is a new ostomy appliance developed by Coloplast A/S
  Arms: Coloplast Test C , Coloplast Test D, Own product
Device: Coloplast Test D — Coloplast Test D is a new ostomy appliance developed by Coloplast A/S
  Arms: Coloplast Test C , Coloplast Test D, Own product

SUMMARY:
To assess the functionality and safety of the test products and also assess the products ability to collect stool without interfering with the stoma.

ELIGIBILITY:
Inclusion Criteria:

1. Had given written informed consent
2. Was at least 18 years of age
3. Was able to handle the appliances themselves or with help from a caregiver (e.g. spouse)
4. Had an ileostomy with a diameter between 15-45 mm
5. Have had an ileostomy for at least 3 months
6. Currently used a 2-piece flat appliance

Exclusion Criteria:

1. Used irrigation during the investigation (flush stoma with water)
2. Currently received or had within the past 2 months received radio- and/or chemotherapy.
3. Currently received or had within the past month received local or systemic steroid treatment in the peristomal area.
4. Was pregnant or breast feeding
5. Participated in other interventional studies that could interfere with this one or had previously participated in this investigation.
6. Had a baseplate wear time of more than three days
7. Suffered from peristomal skin problems that precluded participation in the investigation (assessed by the investigation nurse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Birte p Jakobsen, MD, Principal Investigator — Medical director

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subject were recruited through the Danish Coloplast user data base.
Pre-assignment Details: 28 subjects were randomized. However 2 subject were wrongly randomized. 1 subject was allocated to test Test D in the First period,1 subject First tested Test A followed by Test D.
  Two subject discontinued the testing of the new test products collected data on own product.
  These factors disturb the participant flow chart.
Groups:
- Coloplast Test D, Coloplast Test C, Own Product: The subjects first test Coloplast Test D and thereafter Coloplast Test C and finally their own product for 14 days
  Coloplast Test D: Coloplast Test A is a new ostomy appliance developed by Coloplast A/S
  Coloplast Test C: Coloplast Test B is a newly developed ostomy appliance developed by Coloplast A/S
  Own product: Own product is tested to get baseline results. Own product can be any 2-piece product that is commercially available. The manufactures can be Coloplast, Hollister, Convatec, Dansac, B. Braun and others.
- Oloplast Test A, Coloplast Test D, Own Product: The subjects first test Coloplast Test A and thereafter Coloplast Test D and finally their own product for 14 days
  Coloplast Test A: Coloplast Test A is a new ostomy appliance developed by Coloplast A/S
  Coloplast Test D: Coloplast Test D is a newly developed ostomy appliance developed by Coloplast A/S
  Own product: Own product is tested to get baseline results. Own product can be any 2-piece product that is commercially available. The manufactures can be Coloplast, Hollister, Convatec, Dansac, B. Braun and others.
Period: First Test Period (Test A or Test C)
Arm/Group | Coloplast Test A, Coloplast Test B, Own Product | Coloplast Test C , Coloplast Test D, Own Product | Coloplast Test D, Coloplast Test C, Own Product | Oloplast Test A, Coloplast Test D, Own Product
Started | 14 | 12 | 1 | 1
Completed | 7 | 8 | 0 | 1
Not Completed | 7 | 4 | 1 | 0
Not completed — Lack of Efficacy | 5 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0
Period: Second Test Period (Test B or Test D)
Arm/Group | Coloplast Test A, Coloplast Test B, Own Product | Coloplast Test C , Coloplast Test D, Own Product | Coloplast Test D, Coloplast Test C, Own Product | Oloplast Test A, Coloplast Test D, Own Product
Started | 7 | 8 | 0 | 1
Completed | 6 | 7 | 0 | 1
Not Completed | 1 | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0 | 0
Period: Third Test Period (Own Product)
Arm/Group | Coloplast Test A, Coloplast Test B, Own Product | Coloplast Test C , Coloplast Test D, Own Product | Coloplast Test D, Coloplast Test C, Own Product | Oloplast Test A, Coloplast Test D, Own Product
Started | 8 (One subject who discontinued testing Test A proceeded to test Own product afterwards.) | 8 (One subject who discontinued testing Test C proceeded to test Own product afterwards) | 0 | 1
Completed | 8 | 8 | 0 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study Population
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Degree of Leakage
Description: Degree of leakage is measured on a 24 point scale where 0 represents no leakage (best possible outcome) and 24 represents leakage on the whole plate (worst possible outcome).
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: baseplates
Groups:
- Coloplast Test A: Subjects testing Test A
- Coloplast Test B: Subjects testing Test B
- Coloplast Test C: Subjects testing Test C
- Coloplast Test D: Subjects testing Test D
- Own Product: Subjects collecting data on own product
Arm/Group | Coloplast Test A | Coloplast Test B | Coloplast Test C | Coloplast Test D | Own Product
Number analyzed (Participants) | 15 | 7 | 12 | 10 | 16
Number analyzed (baseplates) | 85 | 43 | 72 | 61 | 87
units on a scale | 6.4 (5.5) | 3.4 (4.2) | 7.0 (4.7) | 7.0 (4.0) | 1.9 (3.1)

ADVERSE EVENTS:
Description: 15 A=14 Coloplast TestA, Coloplast TestB..+1 Oloplast TestA, Coloplast TestD.. 7 B=7 Coloplast TestA, Coloplast TestB..(2nd period) 12 C=12 Coloplast TestC, Coloplast TestD.. 10 D=8 Coloplast TestC, Coloplast TestD..(2nd period)+1 Oloplast Test A, Coloplast Test D..(2nd period)+1 Coloplast Test D..
  16 own product=7 Coloplast Test A, Coloplast Test B..+8 Coloplast Test C, Coloplast Test D..+1 Oloplast Test A, Coloplast Test D..(incl. 2, not completing 2nd period, collecting own product data)
Arm/Group | Coloplast Test A | Coloplast Test B | Coloplast Test C | Coloplast Test D | Own Product
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/7 | 0/12 | 1/10 | 0/16
Other Adverse Events (participants affected / at risk) | 5/15 | 0/7 | 6/12 | 3/10 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coloplast Test A (N=15) | Coloplast Test B (N=7) | Coloplast Test C (N=12) | Coloplast Test D (N=10) | Own Product (N=16)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — The serious adverse event was not related to the investigational device
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coloplast Test A (N=15) | Coloplast Test B (N=7) | Coloplast Test C (N=12) | Coloplast Test D (N=10) | Own Product (N=16)
peristomal skin problem (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0) | 5 (6) | 3 (3) | 0 (0)
Wound peristomal skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Itching peristomal skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes